CLINICAL TRIAL: NCT03634774
Title: CHOICE Plus Program: Supporting Relationship-centred Mealtimes for Long-term Care
Acronym: CHOICE+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Principal Investigator, Heather Keller, Professor, University of Waterloo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ORE22635
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Dementia; Long-term Care
Keywords: meals; staff training
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Step-wedge design; all three groups receive the intervention but two are wait list control for varied amounts of time
Who Masked: Investigator, Outcomes Assessor
Masking Description: Mealtime observations are completed by assessors who are blinded to the order in which sites receive the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Step 1 CHOICE+ (Experimental): Receives the intervention first
  Interventions: Other: CHOICE+ Training Program
- Step 2 CHOICE+ (Other): Received intervention four months after baseline
  Interventions: Other: CHOICE+ Training Program
- Step 3 CHOICE+ (Other): Receives intervention eight months after baseline
  Interventions: Other: CHOICE+ Training Program

INTERVENTIONS:
Other: CHOICE+ Training Program — CHOICE+ is a program where team members and other stakeholders are engaged in making changes to dining in a long term care home to improve the experience. An external coach supports behaviour change.

SUMMARY:
Enhancing the mealtime experience through changing the social and physical aspects of dining holds the potential to not only improve food intake among residents, but enhance their quality of life. The CHOICE+ Program is designed to support relationship-centred mealtimes in long-term care (LTC). This current study will pilot the CHOICE+ Program over the course of 18 months in three LTC homes with the support of a single external facilitator. The research team will collect data at mealtimes and from staff, residents and family members to determine what changes occurred and how this impacted the mealtime experience. The results of this study will provide insight into the efficacy of the CHOICE+ Program and if the program holds potential to improve mealtimes for residents in LTC through relationship-centered dining, as well as capacity building among those who live and work in the home to identify areas for improvement and work together to make change.

DETAILED DESCRIPTION:
This study employs a stepped wedged design that includes three long-term care homes (Site A, Site B, Site C) located within Southern Ontario. Each LTC home will have approximately 12 months to implement the CHOICE+ Program and demonstrate sustainability for the last few weeks; the study will run for 18 months due to the staggered entry of sites into the intervention (Site A: Month 1; Site B: Month 4; Site C: Month 7).

Over the course of 12 months for each Site, the CHOICE+ Program components will be delivered to a single care unit using a 4-phase approach. Transitions from one phase to the next will be entirely dependent upon the context and readiness of those participants involved in the study (i.e., timing between phases may differ amongst LTC homes). A single external facilitator from the University of Waterloo will lead this implementation process. The principal investigator (PI; H. Keller) will assist in guiding the external facilitator through the implementation process and support debriefing sessions. A blinded trained assessor will conduct mealtime experience audits (Mealtime Scan Plus) every 12 weeks starting at Month 1 for Sites A, B, and C, regardless of the implementation start times (i.e., Site A at Month 1; Site B and Month 4; Site C and Month 7). A physical dining room audit will be conducted at four time points (Dining Environment Audit Protocol). Staff, resident and family/volunteer dining experience questionnaires will be completed at four time points as well. Below is sequential description of the implementation process of the CHOICE+ Program in a single site, while accounting for pre-implementation activities:

PHASE 1: PRE-DEVELOPMENT (Week 0)

- PI and facilitator meets with LTC home management/administrators (i.e., Unit Care Coordinators (UCC), Director of Food Service (DFS), Registered Dietitian (RD), and General Manager (GM)) to describe purpose of CHOICE+ Program, address questions and ensure commitment. Once roles and responsibilities are discussed and agreed upon, the researchers will tour the care unit to obtain an understanding of specific contextual factors. A CHOICE+ Newsletter item for residents, family, and volunteers will be distributed to raise awareness of the program. A CHOICE+ Information Letter will be distributed to all staff members, posters with information session dates and times will be posted, and information brochures will be available around the care unit for care staff, residents, family members, and volunteers.

PHASE 2: DEVELOPMENT (Week 1 - Week 8)

* Weeks 1-2: In-services and/or informal connections made by the external facilitator to raise awareness and promote the CHOICE+ Program among care staff, residents, family members, and volunteers on the care unit. Feedback and knowledge exchange with care unit will be sought during these information sessions to gain contextual understanding of specific needs of that care unit's mealtimes.

  * MTS+ Audit 1 data collection by assessor using Mealtime Scan for Long-Term Care PLUS (MTS+), a validated tool to assess the psychosocial and physical environments of a mealtime. Prior to the start of MTS+ Data Collection, posters notifying residents, staff, family members, and volunteers that observations are taking place will be posted in the dining areas.
  * The Dining Environment Audit Protocol (DEAP) is completed when the dining room is empty.
* Week 3: CHOICE+ Dining Team (CDT) that includes residents, family members, care staff (minimum 2), volunteers (if available on unit), and management (minimum 1) will be formed to work closely with external facilitator and care unit to identify aspects of mealtimes that need improvement and support. Two Mealtime Champions (MT Champions) will be identified by the group and/or management as leaders and will act as the key contacts for the facilitator. As part of the team building process and to raise awareness, the CDT will complete a questionnaire about their organization's readiness to make change. As this is a change management step, an information letter and consent for will not be used. The Team Mealtime Experience Questionnaire (TMEQ) will be administered by the facilitator to participating care staff to reflect upon their role in the dining room during meals after informed written consent is provided. Residents, family members, and volunteers will have the option of completing a Dining Experience Questionnaire (DEQ) to share their feelings about mealtimes on the care unit. A separate questionnaire will be available for residents and family members/volunteers and informed written consent or assent in the event the resident is unable to sign a consent form will be provided.
* Weeks 4-8: Training and equipping the CDT on CHOICE+ Principles and change management approaches will take place over 4 meetings hosted by the external facilitator. The themes of these meetings include Meeting #1: CDT Role and CHOICE+ Program overview; Meeting #2: CHOICE+ Education Modules; Meeting #3: Feedback of Audit 1 MTS+, TMEQ, DEAP, and DEQ results. Results will be shared first with the CDT then with the rest of the care unit for review and reflection using the most appropriate communication methods identified by the CDT (i.e., bulletin boards, huddles, posters, etc.); and Meeting #4: Process of making change and priority setting.

PHASE 3: INTENSIVE (Weeks 9-36)

* Weeks 9-10: All care staff on the unit and those residents and family members who are interested in participating in CHOICE+, in addition to the CDT, will complete the CHOICE+ Education Modules (mobile based short videos). In situations where there are new members of the care unit (i.e., care staff, residents and their family members) will also be provided with this education.
* Weeks 9-12: CDT engages with broader care unit to share Audit 1 MTS+, DEAP, TMEQ, and DEQ results to obtain feedback. Communication methods that are most suited to the care unit, for example, posters, meetings, bulletin boards, etc., will be used to share these audit findings. The CDT will engage with the broader care unit to select those mealtime areas for improvement that are most important to neighbours, care staff, and family members.
* Weeks 12-36: The CDT will take these priority areas and work as a team to identify how to make changes and improvements using a variety of behaviour change techniques using a Plan-Do-Study-Act (PDSA) cycle framework. Once a practice change is becoming embedded, a new priority for improvement will be worked through by the CDT and PDSA cycles used to test the improvement. The CDT will be responsible for on-going monitoring of the PDSA cycles in the care unit with support from the facilitator until Week 36 where the facilitator will then begin to reduce their role and the CDT will take on full leadership of the changes being made on the care unit.
* Data collection will using the TMEQ, MTS+, DEAP, and DEQ will follow a schedule for all three sites (see below in "Data Collection") with results fed back to the CDT and the unit team to support change in practice. Mealtime Practices Checklist and Dining Room Checklist will be used as change management activities and self-reflection by the CDT and unit team. As use of these checklists is part of the change process directed by the CDT, informed consent will not be used prior to completion and if forms are collected they will be anonymous for summarization and discussion.

PHASE 4: SUSTAINING (WEEKS 37-52)

* Week 37-52: The sustaining phase will involve ensuring that any new care staff, residents and their family members have access to the CHOICE+ Education Modules. CDT will continue to work the process of change by identifying what needs to improve, how to make the change and completing small tests with PDSA cycles to work through the improvement or new process. DEAP, MTS+, TMEQ, and DEQ results will continue to be provided to the CDT to support change practices and they will continue to use the Mealtime Practices Checklist and other informal self-monitoring data to embed changes. The CDT will continue to hold weekly meetings to monitor the progress of the PDSA cycles and make any necessary modifications to the action plan or its implementation strategies. The facilitator will help the CDT to develop a sustainability plan for the CHOICE+ Program, after which the facilitator will remove herself from the care unit and limit communication either via phone or email with the CDT.
* Data collection will using TMEQ, MTS+, DEAP, and DEQ will follow a schedule for all three sites (see below) with results fed back to the CDT and the unit tem to support change in practice. Mealtime Practices Checklist and Dining Room Checklist will be used as change management activities and self-reflection by the CDT and unit team.
* Week 48-52: External facilitator will complete key informant semi-structured interviews with CDT members including care staff home management residents family members), and volunteers on the CHOICE+ program. It is anticipated than between 10-15 interviews will be conducted at each site. Standard informed consent/assent process will be followed for each potential interview participant.

ELIGIBILITY:
Inclusion Criteria:

* Residents living in the CHOICE+ study units at three long-term care homes in South-Western Ontario

Exclusion Criteria:

* Residents who do not live in the chosen area for these homes, or live in different homes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Mealtime Scan | 16 months
  Observational instrument that objectively measures the mealtime experience

SECONDARY OUTCOMES:
Team member Mealtime Experience | Before /after 12 months of intervention
  This 23 item questionnaire rates team member experience with dining
Resident/Family member dining quality | Baseline/after 12 months of intervention
  This five item questionnare provides the perspective of residents and family on the dining experience

CONTACTS AND LOCATIONS:
Overall Officials: Heather Keller, PhD, Principal Investigator — University of Waterloo
Locations (3):
- Canada (3):
  - Erin Mills Lodge, Mississauga
  - Extendicare Bayview, North York
  - Christie Gardens, Toronto

IPD SHARING:
Plan to Share IPD: No